CLINICAL TRIAL: NCT05903170
Title: A Randomised Trial of Shock Energy for Electrical Cardioversion of Persistent Atrial Fibrillation
Brief Title: Shock Energy for Electrical Cardioversion of Persistent Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wellington Hospital (Other Government)
Responsible Party: Principal Investigator, Allan Plant, Principal Investigator, Wellington Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRH DCCV
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Defibrillators

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to undergo cardioversion with one of two defibrillators at either 200J or 360J. Randomization will occur by a random number generator, and the chance of being in either arm is 50%.
  Participants in each arm will undergo up to three shocks at the energy-level to which they have been randomized, using a standardized procedure. For participants randomized to the lower energy level who fail to return to normal rhythm after three shocks, they will be given a fourth shock at the higher energy level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 360J LifePak Monitor/Defibrillator (Active Comparator): The standardised cardioversion protocol below performed with a 360J shock from a Lifepak Monitor/Defibrillator.
  1. First shock with anteroposterior pad configuration
  2. In event of failure of the above, a second shock with anterolateral pad configuration
  3. In event of failure of the above, a third shock with anteroposterior pad configuration + manual pad pressure
  Interventions: Device: 360J LifePak Monitor/Defibrillator
- 200J Philips HeartStart MRx Monitor/Defibrillator (Active Comparator): The standardised cardioversion protocol below performed with a 200J shock from a Philips HeartStart MRx Monitor/Defibrillator.
  1. First shock with anteroposterior pad configuration
  2. In event of failure of the above, a second shock with anterolateral pad configuration
  3. In event of failure of the above, a third shock with anteroposterior pad configuration + manual pad pressure
  4. The addition of a fourth 'rescue' shock at 360J using the LifePak Monitor/Defibrillator with pads in the anteroposterior configuration in the event of the first three steps failing to cardiovert to sinus rhythm
  Interventions: Device: 200J Philips HeartStart MRx Monitor/Defibrillator

INTERVENTIONS:
Device: 360J LifePak Monitor/Defibrillator — The LifePak Monitor/Defibrillator is a commonly-used defibrillator in New Zealand hospitals for cardioverting atrial fibrillation. It delivers a biphasic waveform shock with a titratable maximum energy of 360J.
  Arms: 360J LifePak Monitor/Defibrillator
Device: 200J Philips HeartStart MRx Monitor/Defibrillator — The Philips HeartStart MRx Monitor/Defibrillator is a commonly-used defibrillator in New Zealand hospitals for cardioverting atrial fibrillation. It delivers a biphasic waveform shock with a titratable maximum energy of 200J.
  Arms: 200J Philips HeartStart MRx Monitor/Defibrillator

SUMMARY:
The goal of this clinical trial is to compare the efficacy of a maximum output shock for cardioverting atrial fibrillation between two commonly used defibrillators in New Zealand . These machines have different maximum energy outputs, and to date no head-to-head comparison cardioverting atrial fibrillation between the two has been undertaken.

The main question it aims to answer is whether either device is more likely to cardiovert patients referred for atrial fibrillation.

Participants will be randomized to undergo cardioversion with one of two defibrillators at either 200J or 360J. Participants in each arm will undergo up to three shocks at the energy-level to which they have been randomized, using a standardized procedure. For participants randomized to the lower energy level who fail to return to normal rhythm after three shocks, they will be given a fourth shock at the higher energy level.

All participants will then be asked to undertake a blood test the day following the cardioversion, and receive a follow up phone call. These are to ensure there is no difference in the safety of the procedure between the two energy levels. It is worth noting that these two components of the study (the blood test and phone call) are the only additional time commitment that is expected to be involved if you choose to participate in the study.

DETAILED DESCRIPTION:
Atrial fibrillation is the world's most common arrhythmia, with an incidence that is increasing in Western countries. One-in-four adults will experience atrial fibrillation at some point in their life.

Strategies for the management of atrial fibrillation include rate control, prophylaxis against stroke, lifestyle modification, and restoration of sinus rhythm through medical or electrical cardioversion. Electrical cardioversion for the restoration of sinus rhythm was first described by Lown and colleagues in 1962, and has undergone a number of procedural advances in the intervening six decades. Chief amongst these was a transition from cardioverting using monophasic to biphasic waveforms, something unequivocally demonstrated to increase cardioversion success, with lower energy, current, and less skin and muscle damage than monophasic devices. Yet the majority of the data which continues to guide cardioversion is derived from the era of monophasic therapy.

Data from cardioversion with monophasic waveforms suggests that the use of higher initial shock energy is associated with higher first shock success, fewer shocks, and lower levels of skeletal muscle injury, with no increase in troponin to suggest greater cardiac injury. Likewise, studies of shock energy using biphasic devices have demonstrated benefit of maximum fixed shock energy. However, whilst the energy of a defibrillator remains entrenched in the descriptive vocabulary of cardioversion for atrial fibrillation, it is the flow of current across the myocardium that achieves cardioversion, and resuscitation guidelines have previously recommended a switch to the more physiologic current-based description.

Different defibrillators deliver different currents at the same energy setting based on the capacitance of the device. As such, manufacturers of defibrillators recommend different energy levels for cardioverting atrial fibrillation with some standard biphasic defibrillators (Philips HeartStart MRx Monitor/Defibrillator) unable to deliver higher than 200J energy, while some (Lifepak 15 Monitor/Defibrillator) extend to 360J. No studies have compared initial 200J vs. 360J shock energies between these devices for cardioverting persistent atrial fibrillation.

This study is a single centre randomized non-blinded study of the effectiveness of 200J vs. 360J fixed output biphasic electrical cardioversion in patients undergoing electrical cardioversion of persistent atrial fibrillation. The study hypothesis is that cardioversion with shock energy fixed to 360J delivered by a LifePak Monitor/Defibrillator is more efficacious than a 200J delivered by a Philips HeartStart MRx Monitor/Defibrillator, without worsening safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patients undergoing either elective outpatient or non-emergent inpatient cardioversion for atrial fibrillation
* Eligible for anticoagulation
* Reliably anticoagulated for ≥three weeks prior to cardioversion, AF onset within 48hrs of cardioversion, or left atrial thrombus excluded on transoesophageal echocardiogram
* Able to consent to cardioversion, and study participation

Exclusion Criteria:

* Contraindication to anticoagulation
* Atrial flutter
* Emergent cardioversion
* Implantable cardiac device (PPM or ICD)
* Unable to consent to cardioversion and/or study participation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Cardioversion efficacy | During Procedure (1 Hour)
  Percentage of patients successfully cardioverted to sinus rhythm

SECONDARY OUTCOMES:
Shock number | During Procedure (1 Hour)
  Number of shocks required to cardiovert to sinus rhythm
Cumulative energy | During Procedure (1 Hour)
  Total energy delivered during procedure

OTHER OUTCOMES:
Safety outcome: skin erythema | 2 hours after procedure
  Proportion of patients with documented skin erythema at discharge
Safety outcome: pain score | 2 hours after procedure
  Average pain score on a 10 point numerical rating scale from 0 (no pain) to 10 (severe pain)
Safety outcome: troponin elevation | 24 hours after procedure
  Proportion of patients with a significant troponin elevation (defined as a troponin greater the ULN and ≥50% increase from baseline)
Safety outcome: troponin change from baseline | 24 hours after procedure
  Average change in troponin from baseline
Safety outcome: creatine kinase change from baseline | 24 hours after procedure
  Average change in creatinine kinase from baseline
Safety outcome: other | 2 hours after procedure
  Any other clinically-significant event requiring change in management (need for temporary pacing / BP support / admission due to complications)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Plant, FRACP, Principal Investigator — Wellington Hospital
Locations (1):
- Wellington Regional Hospital, Wellington, Wellington Region, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boos C, Thomas MD, Jones A, Clarke E, Wilbourne G, More RS. Higher energy monophasic DC cardioversion for persistent atrial fibrillation: is it time to start at 360 joules? Ann Noninvasive Electrocardiol. 2003 Apr;8(2):121-6. doi: 10.1046/j.1542-474x.2003.08205.x. PMID 12848792
- [Background] ECC Committee, Subcommittees and Task Forces of the American Heart Association. 2005 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2005 Dec 13;112(24 Suppl):IV1-203. doi: 10.1161/CIRCULATIONAHA.105.166550. Epub 2005 Nov 28. No abstract available. PMID 16314375
- [Background] Lippi G, Sanchis-Gomar F, Cervellin G. Global epidemiology of atrial fibrillation: An increasing epidemic and public health challenge. Int J Stroke. 2021 Feb;16(2):217-221. doi: 10.1177/1747493019897870. Epub 2020 Jan 19. PMID 31955707
- [Background] Joglar JA, Hamdan MH, Ramaswamy K, Zagrodzky JD, Sheehan CJ, Nelson LL, Andrews TC, Page RL. Initial energy for elective external cardioversion of persistent atrial fibrillation. Am J Cardiol. 2000 Aug 1;86(3):348-50. doi: 10.1016/s0002-9149(00)00932-2. PMID 10922451
- [Background] Koster RW, Dorian P, Chapman FW, Schmitt PW, O'Grady SG, Walker RG. A randomized trial comparing monophasic and biphasic waveform shocks for external cardioversion of atrial fibrillation. Am Heart J. 2004 May;147(5):e20. doi: 10.1016/j.ahj.2003.10.049. PMID 15131555
- [Background] Page RL, Kerber RE, Russell JK, Trouton T, Waktare J, Gallik D, Olgin JE, Ricard P, Dalzell GW, Reddy R, Lazzara R, Lee K, Carlson M, Halperin B, Bardy GH; BiCard Investigators. Biphasic versus monophasic shock waveform for conversion of atrial fibrillation: the results of an international randomized, double-blind multicenter trial. J Am Coll Cardiol. 2002 Jun 19;39(12):1956-63. doi: 10.1016/s0735-1097(02)01898-3. PMID 12084594
- [Background] Schmidt AS, Lauridsen KG, Torp P, Bach LF, Rickers H, Lofgren B. Maximum-fixed energy shocks for cardioverting atrial fibrillation. Eur Heart J. 2020 Feb 1;41(5):626-631. doi: 10.1093/eurheartj/ehz585. PMID 31504412
- [Background] Staerk L, Wang B, Preis SR, Larson MG, Lubitz SA, Ellinor PT, McManus DD, Ko D, Weng LC, Lunetta KL, Frost L, Benjamin EJ, Trinquart L. Lifetime risk of atrial fibrillation according to optimal, borderline, or elevated levels of risk factors: cohort study based on longitudinal data from the Framingham Heart Study. BMJ. 2018 Apr 26;361:k1453. doi: 10.1136/bmj.k1453. PMID 29699974